CLINICAL TRIAL: NCT00644826
Title: Growing Old at Home - Effectiveness and Cost-effectiveness of Preventive Home Visits to Reduce Nursing Home Admissions in the Elderly
Brief Title: Growing Old at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Prof. Dr. phil habil Johann Behrens, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PfVMS-T5
Record Dates: First submitted 2008-03-26; First posted 2008-03-27 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-01

CONDITIONS: Aging
Keywords: randomized controlled trial; public health; Preventive Health Services
MeSH Terms: interventions — Geriatric Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: preventive home visit
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: preventive home visit — A multidimensional geriatric assessment within the dimensions: cognition, health related functioning, risk of falling, nutritional status, social situation, economic situation, mood. Two more home visits: (1) home counseling visit 2-3 weeks after assessment (2) booster session 1 month after home counseling visit
  Other Names: geriatric assessment
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether preventive home visits for people aged 80 and over are effective in the prevention of nursing home admission in Germany.

DETAILED DESCRIPTION:
Regarding demographic changes in Germany it can be assumed that the number of elderly and the resulting need for long term care is increasing in the near future. It is not only an individual's interest but also of public concern to avoid a nursing home admission. Current evidence indicates that preventive home visits can be an effective way to reduce the admission rate in this way making it possible for elderly people to stay longer at home than without home visits. As the effectiveness and cost-effectiveness of preventive home visits strongly depends on existing services in the social and health system existing international results cannot be merely transferred to Germany. Therefore it is necessary to investigate the effectiveness and cost-effectiveness of such an intervention by a randomized controlled trial in Germany.

ELIGIBILITY:
Inclusion Criteria:

* older than 80
* fluent German speaker
* resident of Leipzig or Halle
* living at home (i.e. no nursing home resident)

Exclusion Criteria:

* cognitive impairment
* not able to give informed consent
* care level higher than 1 according to German long term care insurance

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 336 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
nursing home admission rate | 18 months

SECONDARY OUTCOMES:
health care service utilization and costs | 18 months
incremental cost-effectiveness and cost- utility ratio | 18 months
health related functioning | 18 months
health related quality of life | 18 months
prevalence of falls | 18 months
time to nursing home admission | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Johann Behrens, PhD, Principal Investigator — Martin-Luther-Universität Halle-Wittenberg; Steffi Riedel-Heller, MD, Principal Investigator — Universität Leipzig
Locations (2):
- Germany (2):
  - Institut für Gesundheits- und Pflegewissenschaft, Medizinische Fakultät, Martin-Luther-Universität Halle-Wittenberg, Halle, SAN
  - Klinik und Poliklinik für Psychiatrie, Universitätsklinikum Leipzig AöR, Leipzig, SA

REFERENCES:
- [Derived] Brettschneider C, Luck T, Fleischer S, Roling G, Beutner K, Luppa M, Behrens J, Riedel-Heller SG, Konig HH. Cost-utility analysis of a preventive home visit program for older adults in Germany. BMC Health Serv Res. 2015 Apr 3;15:141. doi: 10.1186/s12913-015-0817-0. PMID 25884452
- [Derived] Fleischer S, Roling G, Beutner K, Hanns S, Behrens J, Luck T, Kuske B, Angermeyer MC, Riedel-Heller SG, Heinrich S, Konig HH, Lautenschlager C. Growing old at home - a randomized controlled trial to investigate the effectiveness and cost-effectiveness of preventive home visits to reduce nursing home admissions: study protocol [NCT00644826]. BMC Public Health. 2008 May 28;8:185. doi: 10.1186/1471-2458-8-185. PMID 18507840